CLINICAL TRIAL: NCT03177603
Title: An Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of GSK2586881 in Participants With Pulmonary Arterial Hypertension
Brief Title: A Dose-escalation Study in Subjects With Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206246; 2017-000212-41 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension; Dose-escalation; Safety; Tolerability; GSK2586881
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — alunacedase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GSK2586881 - 0.1 mg/kg (Experimental): Eligible subjects will receive a single dose of 0.1 mg/kg GSK2586881. Dose escalation up to maximum dose of 0.8 mg/kg will occur after 4 subjects have been dosed per cohort and review of safety, tolerability, PK and hemodynamic data up to 24 hours post dose has taken place.
  Interventions: Drug: GSK2586881
- GSK2586881 - 0.2 mg/kg (Experimental): Eligible subjects will receive a single dose 0.2 mg/kg of GSK2586881 IV infusion. Dose escalation up to maximum dose of 0.8 mg/kg will occur after 4 subjects have been dosed per cohort and review of safety, tolerability, PK and hemodynamic data up to 24 hours post dose has taken place.
  Interventions: Drug: GSK2586881
- GSK2586881 - 0.4 mg/kg (Experimental): Eligible subjects will receive a single dose of 0.4 mg/kg of GSK2586881 IV infusion. Dose escalation up to maximum dose of 0.8 mg/kg will occur after 4 subjects have been dosed per cohort and review of safety, tolerability, PK and hemodynamic data up to 24 hours post dose has taken place.
  Interventions: Drug: GSK2586881
- GSK2586881 - 0.8 mg/kg (Experimental): Eligible subjects will receive single dose of 0.8 mg/kg of GSK2586881 IV infusion. Dose escalation will occur after 4 subjects have been dosed per cohort and review of safety, tolerability, PK and hemodynamic data up to 24 hours post dose has taken place.
  Interventions: Drug: GSK2586881

INTERVENTIONS:
Drug: GSK2586881 — GSK2586881 is a clear colorless liquid for IV infusion over 3- 5 minutes and will be administered a maximum dose of 0.8 mg/kg.

SUMMARY:
GSK2586881, a purified intravenous (IV) formulation of soluble recombinant human Angiotensin Converting Enzyme (rhACE2) is being investigated as a treatment for PAH. This GlaxoSmithKline (GSK) study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GSK2586881 in subjects with PAH. This open-label, dose-escalation study will comprise of 4 separate groups based on the planned dose range, and subjects in each group will be administered a single dose of GSK2586881 ranging between 0.1, 0.2, 0.4 and 0.8 milligram per kilogram (mg/kg) via IV route. Dose escalation will occur after 4 subjects have been dosed per cohort and review of safety, tolerability, PK and hemodynamic data up to 24 hours post dose has taken place. A maximum of 27 subjects will be included in the study and the total duration of the study will be up to a maximum of 59 days.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be between 18-75 years of age (inclusive), at the time of signing the informed consent.
* Documented diagnosis of PAH, defined as mPAP > 25 millimeter of mercury (mmHg) and pulmonary wedge pressure (PWP) <= 15.
* Idiopathic PAH (IPAH), Hereditary PAH (HPAH), or PAH associated with collagen vascular disease, or appetite suppressant use.
* World Health Organization (WHO) functional class I, II, or III, stable for at least 8 weeks prior to enrollment.
* Hemodynamically stable on background therapy with no evidence of uncontrolled right heart failure (historic data), as determined by the investigator.
* Six minute walk (6MW) distance, as performed at screening or within 6 months prior to screening, of >= 100 meters (m) and <= 500 m.
* Mean BP of >60 mmHg.
* Receiving stable doses of one or more medications that are approved for treatment of PAH, including endothelin receptor antagonists, phosphodiesterase 5 inhibitors, and/or prostanoids/prostacyclin receptor agonists, for a minimum of 12 consecutive weeks before enrollment.
* Diuretic dose stable for 8 weeks.
* Body weight <= 100 kg and body mass index (BMI) within the range 18-35 kg per m square (kg/m^2) (inclusive).
* Male and/or female (following confirmation of negative pregnancy test for Women of Childbearing Potential [WOCBP]). Women who are pregnant or breastfeeding are excluded.
* Capable of giving signed informed consent.

Exclusion Criteria

* History of systemic hypotension, defined as systolic BP <90 mmHg and/or diastolic BP <50 mmHg.
* Hospitalization for PAH associated deterioration in the previous 6 months.
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance, including all prescribed evaluations and follow-up activities. Concurrent disease or condition that may interfere with study participation or safety include bleeding disorders, arrhythmia, organ transplant, organ failure, current neoplasm, poorly controlled diabetes mellitus, and serious neurological disorders.
* Complex repaired and unrepaired congenital heart disease.
* Subjects with Eisenmenger physiology.
* Alanine transferase (ALT) >2x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Estimated glomerular-filtration-rate (eGFR) <45 milliliter per minute per 1.73 meter square (mL/min/1.73m^2).
* QTc >480 millisecond (msec) or QTc > 500 msec in subjects with bundle branch block.
* Any bleeding concerns as evidenced by International normalized ratio (INR) >1.5 (in subjects not receiving anticoagulation therapy) or platelet count <80,000.
* Hemoglobin (Hb) <10 gram per deciliter (g/dL).
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates participation in the study.
* Any use of an Angiotensin-converting enzyme (ACE) inhibitor or Angiotensin receptor blocker or renin inhibitors within 14 days prior to dosing. Therapy can be stopped to enable inclusion if deemed safe by the subject's treating physician.
* Use of any investigational product (IP) or device within 30 days prior to dosing, or known requirement for any investigational agent prior to completion of all scheduled study assessments.
* Positive human immunodeficiency virus (HIV) antibody test.
* Presence of Hepatitis B surface antigen (HBsAg) at screening.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to starting study treatment.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Participation in the study would result in loss of blood or blood products in excess of 300mL within 65 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* A known or suspected history of alcohol or drug abuse within the 2 years prior to screening.
* Unable to refrain from smoking during the in-house treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (2):
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
- Germany (4):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 2a, open-label, dose-escalation study comprised of 4 cohorts. Participants received GSK2586881 by single intravenous (IV) infusion at following doses: 0.1 milligram per kilogram (mg/kg) or 0.2 mg/kg or 0.4 mg/kg or 0.8 mg/kg.
Pre-assignment Details: A total of 31 participants were screened and of them 7 participants were screen failures and one withdrew consent before dosing. Hence, a total of 23 participants received study treatment. This study was conducted at 4 centers in Germany, 2 centers in Spain, and 2 centers in the United States.
Groups:
- GSK2586881 0.1 mg/kg: Participants received a single IV dose of 0.1 mg/kg GSK2586881 and were followed up till 28 days post-dose.
- GSK2586881 0.2 mg/kg: Participants received a single IV dose of 0.2 mg/kg GSK2586881 and were followed up till 28 days post-dose.
- GSK2586881 0.4 mg/kg: Participants received a single IV dose of 0.4 mg/kg GSK2586881 and were followed up till 28 days post-dose.
- GSK2586881 0.8 mg/kg: Participants received a single IV dose of 0.8 mg/kg GSK2586881 and were followed up till 28 days post-dose.
Period: Cohort 1: Dose Level 0.1 mg/kg (28 Days)
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Started | 4 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2: Dose Level 0.2 mg/kg (28 Days)
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Started | 0 | 5 | 0 | 0
Completed | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 3: Dose Level 0.4 mg/kg (28 Days)
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Started | 0 | 0 | 6 | 0
Completed | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 4: Dose Level 0.8 mg/kg (28 Days)
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Started | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg | Total
Number analyzed (Participants) | 4 | 5 | 6 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.0 (4.97) | 55.4 (14.96) | 52.5 (8.67) | 50.3 (13.35) | 48.8 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 5 | 15
  Male | 1 | 2 | 2 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1 | 1 | 3
  White - White/Caucasian/European Heritage | 4 | 4 | 5 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR)
Description: PVR is the resistance generated by pulmonary circulation. Pulmonary arterial catheters were placed in participants and PVR values were recorded from the right heart catheterization. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: Evaluable Population comprised of all participants who were in the safety population, who completed all Day 1 assessments (including up to 24 hours post dose) and were not deemed to have had major protocol deviations. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  1 hour post-dose (Day 1) | 0.936 [0.725 to 1.208] | 0.885 [0.686 to 1.141] | 0.813 [0.561 to 1.178] | 1.017 [0.862 to 1.198]
  2 hours post-dose (Day 1) | 0.926 [0.671 to 1.279] | 1.043 [0.910 to 1.195] | 0.945 [0.788 to 1.134] | 0.974 [0.823 to 1.153]
  4 hours post-dose (Day 1) | 0.907 [0.552 to 1.490] | 0.895 [0.668 to 1.199] | 0.924 [0.589 to 1.448] | 1.116 [1.050 to 1.186]

2. Primary Outcome: Change From Baseline in Cardiac Output (CO)
Description: CO is the amount of blood pumped by the heart per minute. Pulmonary arterial catheters were placed in participants and CO values were recorded from the right heart catheterization. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  1 hour post-dose (Day 1) | 1.046 [0.881 to 1.240] | 1.079 [0.966 to 1.206] | 1.076 [0.758 to 1.528] | 0.990 [0.948 to 1.033]
  2 hours post-dose (Day 1) | 1.025 [0.829 to 1.269] | 1.029 [0.950 to 1.116] | 0.929 [0.712 to 1.210] | 1.012 [0.944 to 1.085]
  4 hours post-dose (Day 1) | 1.114 [0.804 to 1.545] | 1.138 [0.949 to 1.365] | 0.882 [0.734 to 1.060] | 1.002 [0.935 to 1.075]

3. Primary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (mPAP)
Description: The pulmonary artery pressure is a measure of the blood pressure found in the main pulmonary artery. Pulmonary arterial catheters were placed in participants and mPAP values were recorded from the right heart catheterization. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  1 hour post-dose (Day 1) | 0.950 [0.781 to 1.154] | 0.995 [0.960 to 1.032] | 0.939 [0.799 to 1.104] | 0.989 [0.879 to 1.114]
  2 hours post-dose (Day 1) | 0.937 [0.781 to 1.126] | 0.994 [0.924 to 1.070] | 0.910 [0.766 to 1.081] | 0.996 [0.867 to 1.144]
  4 hours post-dose (Day 1) | 0.991 [0.812 to 1.211] | 1.029 [0.881 to 1.202] | 0.973 [0.897 to 1.054] | 1.062 [0.958 to 1.177]

4. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment.
Time Frame: Up to Day 28
Population: Safety Population comprised of all participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Participants | 1 | 3 | 5 | 2

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Any untoward event resulting in death, life threatening, requiring hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention were categorized as SAE.
Time Frame: Up to Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alkaline Phosphatase, Alanine Amino Transferase and Aspartate Amino Transferase
Description: Blood samples were collected for the assessment of clinical chemistry parameters: alkaline phosphatase, alanine amino transferase (ALT) and aspartate amino transferase (AST). Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
International units per liter
  Alkaline phosphatase, 24 hours post-dose (Day 1) | 4.8 (8.42) | -1.4 (7.44) | 5.3 (3.08) | 3.1 (3.48)
  Alkaline phosphatase, Day 7 to Day 14 | 6.5 (5.00) | 3.2 (4.21) | 3.0 (3.52) | 2.6 (4.31)
  ALT, 24 hours post-dose (Day 1) | -2.0 (2.16) | 0.0 (1.58) | -1.8 (3.76) | -0.1 (2.17)
  ALT, Day 7 to Day 14 | 1.3 (0.96) | 1.8 (3.27) | -4.3 (12.94) | 0.9 (4.85)
  AST, 24 hours post-dose (Day 1) | 0.0 (1.63) | -0.4 (0.55) | 0.5 (1.76) | -1.8 (3.77)
  AST, Day 7 to Day 14 | 2.8 (2.50) | 1.4 (1.67) | -0.3 (3.67) | -0.9 (6.71)

7. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Creatinine
Description: Blood samples were collected for the assessment of clinical chemistry parameters: direct bilirubin, total bilirubin and creatinine. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Micromoles per liter
  Direct bilirubin, 24 hours post-dose (Day 1) | 2.0 (1.63) | 0.4 (0.89) | 0.3 (1.97) | 1.0 (2.14)
  Direct bilirubin, Day 7 to Day 14 | 1.0 (1.15) | 0.0 (0.00) | 0.0 (1.26) | 0.5 (2.56)
  Total bilirubin, 24 hours post-dose (Day 1) | 3.0 (4.16) | 0.8 (1.79) | 0.7 (4.84) | 4.8 (6.76)
  Total bilirubin, Day 7 to Day 14 | 1.5 (3.42) | 0.4 (2.61) | -1.7 (3.44) | 0.0 (4.14)
  Creatinine, 24 hours post-dose (Day 1) | 5.08 (4.102) | 10.80 (6.110) | 12.22 (20.214) | 1.76 (2.759)
  Creatinine, Day 7 to Day 14 | -1.12 (6.530) | 8.68 (13.353) | 4.57 (9.638) | 3.20 (4.885)

8. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Blood Urea Nitrogen (BUN)
Description: Blood samples were collected for the assessment of clinical chemistry parameters: calcium, glucose, potassium, sodium and BUN. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Millimoles per liter
  Calcium, 24 hours post-dose (Day 1) | 0.035 (0.1427) | 0.012 (0.0867) | 0.047 (0.1033) | 0.060 (0.0466)
  Calcium, Day 7 to Day 14 | 0.025 (0.1399) | 0.064 (0.0888) | 0.047 (0.1250) | 0.115 (0.0583)
  Glucose, 24 hours post-dose (Day 1) | 0.85 (0.957) | 1.10 (1.398) | 0.50 (1.752) | 0.89 (2.039)
  Glucose, Day 7 to Day 14 | 0.95 (1.760) | -0.32 (0.646) | -0.57 (0.635) | -0.20 (1.995)
  Potassium, 24 hours post-dose (Day 1) | 0.28 (0.377) | 0.18 (0.179) | 0.08 (0.306) | -0.05 (0.239)
  Potassium, Day 7 to Day 14 | 0.10 (0.356) | 0.22 (0.148) | 0.25 (0.207) | 0.18 (0.301)
  Sodium, 24 hours post-dose (Day 1) | -1.3 (1.26) | -0.6 (2.30) | -0.2 (1.47) | -1.0 (1.85)
  Sodium, Day 7 to Day 14 | -0.3 (4.19) | 0.0 (1.87) | 0.5 (1.64) | 0.0 (1.60)
  BUN, 24 hours post-dose (Day 1) | 0.00 (1.080) | -0.20 (0.758) | 0.83 (1.033) | -0.25 (0.463)
  BUN, Day 7 to Day 14 | -0.25 (1.258) | 1.50 (1.541) | 0.00 (1.000) | 0.31 (1.067)

9. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Total Protein
Description: Blood samples were collected for the assessment of clinical chemistry parameter, total protein. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Grams per liter
  24 hours post-dose (Day 1) | 1.3 (6.13) | 0.6 (3.78) | 1.8 (2.93) | 2.6 (3.66)
  Day 7 to Day 14 | 1.5 (2.38) | 6.2 (4.55) | 2.0 (4.73) | 4.9 (3.31)

10. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and White Blood Cell (WBC) Count
Description: Blood samples were collected for the assessment of hematology parameters: basophils, eosinophils, lymphocytes, monocytes, total neutrophils (T.neutrophils), platelet count and WBC count. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Giga cells per liter
  Basophils, 24 hours post-dose (Day 1), n=4,4,6,3: number analyzed (Participants) | 4 | 4 | 6 | 3
  Basophils, 24 hours post-dose (Day 1), n=4,4,6,3 | -0.008 (0.0359) | 0.013 (0.0206) | -0.005 (0.0302) | 0.003 (0.0115)
  Basophils, Day 7 to Day 14, n=4,5,6,8 | 0.000 (0.0327) | 0.002 (0.0192) | 0.008 (0.0306) | 0.003 (0.0238)
  Eosinophils, 24 hours post-dose (Day 1), n=4,4,6,3: number analyzed (Participants) | 4 | 4 | 6 | 3
  Eosinophils, 24 hours post-dose (Day 1), n=4,4,6,3 | 0.007 (0.0695) | 0.018 (0.0222) | 0.012 (0.0662) | -0.007 (0.0503)
  Eosinophils, Day 7 to Day 14, n=4,5,6,8 | -0.035 (0.0835) | 0.004 (0.0230) | -0.025 (0.0807) | 0.023 (0.1004)
  Lymphocytes, 24 hours post-dose (Day 1), n=4,4,6,3: number analyzed (Participants) | 4 | 4 | 6 | 3
  Lymphocytes, 24 hours post-dose (Day 1), n=4,4,6,3 | 0.000 (0.5509) | -0.070 (0.1612) | -0.157 (0.1558) | 0.190 (0.4553)
  Lymphocytes, Day 7 to Day 14, n=4,5,6,8 | -0.025 (0.4277) | -0.054 (0.1422) | -0.250 (0.2001) | 0.130 (0.4032)
  Monocytes, 24 hours post-dose (Day 1), n=4,4,6,3: number analyzed (Participants) | 4 | 4 | 6 | 3
  Monocytes, 24 hours post-dose (Day 1), n=4,4,6,3 | 0.050 (0.0673) | -0.028 (0.0914) | 0.098 (0.1125) | 0.140 (0.0700)
  Monocytes, Day 7 to Day 14, n=4,5,6,8 | 0.038 (0.1066) | 0.038 (0.0998) | 0.047 (0.1263) | 0.091 (0.1654)
  T.neutrophils, 24 hours post-dose(Day1),n=4,4,6,3: number analyzed (Participants) | 4 | 4 | 6 | 3
  T.neutrophils, 24 hours post-dose(Day1),n=4,4,6,3 | 0.643 (1.0052) | 0.415 (0.3924) | 0.738 (0.5615) | 0.727 (0.7298)
  T.neutrophils, Day 7 to Day 14, n=4,5,6,8 | 0.185 (0.9008) | 0.504 (0.4884) | 0.397 (1.3173) | 0.366 (0.7204)
  Platelets, 24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  Platelets, 24 hours post-dose (Day 1), n=4,4,6,5 | 11.8 (36.28) | -33.0 (73.51) | 7.8 (16.65) | 12.6 (27.74)
  Platelets, Day 7 to Day 14, n=4,5,6,8 | 35.3 (17.40) | 19.8 (45.03) | 14.3 (52.89) | 23.4 (24.44)
  WBC count, 24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  WBC count, 24 hours post-dose (Day 1), n=4,4,6,5 | 0.35 (1.330) | 0.30 (0.183) | 0.68 (0.542) | 2.16 (2.492)
  WBC count, Day 7 to Day 14, n=4,5,6,8 | -0.20 (1.334) | 0.46 (0.498) | 0.20 (1.355) | 0.64 (0.588)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the assessment of hematology parameter, hemoglobin. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Grams per liter
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | 1.8 (11.09) | 2.0 (5.72) | 5.0 (4.77) | 3.0 (5.61)
  Day 7 to Day 14, n=4,5,6,8 | -4.3 (6.55) | 3.4 (5.98) | -1.5 (7.09) | 4.0 (5.15)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for the assessment of hematology parameter, hematocrit. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Proportion of red blood cells in blood
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | 0.0030 (0.02858) | 0.0053 (0.02156) | 0.0098 (0.01546) | 0.0140 (0.02448)
  Day 7 to Day 14, n=4,5,6,8 | -0.0225 (0.00929) | 0.0104 (0.02173) | 0.0030 (0.02391) | 0.0135 (0.01891)

13. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin
Description: Blood samples were collected for the assessment of hematology parameter, mean corpuscle hemoglobin. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Picograms
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | -0.08 (0.150) | 0.05 (0.507) | 0.25 (0.302) | -0.10 (0.235)
  Day 7 to Day 14, n=4,5,6,8 | 0.10 (0.483) | 0.04 (0.182) | -0.33 (0.314) | 0.15 (0.177)

14. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume
Description: Blood samples were collected for the assessment of hematology parameter, mean corpuscle volume. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Femtoliters
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | -0.5 (2.52) | 0.0 (0.82) | -0.5 (0.84) | 0.6 (1.95)
  Day 7 to Day 14, n=4,5,6,8 | -1.5 (2.08) | -0.2 (0.84) | 0.7 (1.03) | 0.8 (1.04)

15. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell (RBC) Count
Description: Blood samples were collected for the assessment of hematology parameter: RBC count. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Trillion cells per liter
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | 0.03 (0.435) | 0.03 (0.287) | 0.13 (0.163) | 0.12 (0.192)
  Day 7 to Day 14, n=4,5,6,8 | -0.20 (0.183) | 0.14 (0.261) | 0.00 (0.310) | 0.11 (0.203)

16. Secondary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes
Description: Blood samples were collected for the assessment of hematology parameter: reticulocytes. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose), 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in blood
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Percentage of reticulocytes in blood
  24 hours post-dose (Day 1), n=4,4,6,5: number analyzed (Participants) | 4 | 4 | 6 | 5
  24 hours post-dose (Day 1), n=4,4,6,5 | 0.0012 (0.00330) | 0.0017 (0.00310) | 0.0017 (0.00216) | 0.0000 (0.00100)
  Day 7 to Day 14, n=4,5,6,8 | 0.0058 (0.00411) | 0.0014 (0.00358) | 0.0025 (0.00333) | 0.0040 (0.00325)

17. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Method
Description: Urine samples were collected to assess urine bilirubin, urine occult blood, urine glucose, urine ketones, and urine protein by dipstick test. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine bilirubin, urine occult blood, urine glucose, urine ketones and urine protein can be read as negative, trace, 1+, 2+ and 3+ indicating proportional concentrations in the urine sample.
Time Frame: 24 hours post-dose (Day 1)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Participants
  Bilirubin, 24 hours post-dose (Day 1), negative | 4 | 5 | 6 | 8
  Bilirubin, 24 hours post-dose (Day 1), trace | 0 | 0 | 0 | 0
  Bilirubin, 24 hours post-dose (Day 1), 1+ | 0 | 0 | 0 | 0
  Bilirubin, 24 hours post-dose (Day 1), 2+ | 0 | 0 | 0 | 0
  Bilirubin, 24 hours post-dose (Day 1), 3+ | 0 | 0 | 0 | 0
  Occult Blood, 24 hours post-dose (Day 1), negative | 2 | 5 | 4 | 7
  Occult Blood, 24 hours post-dose (Day 1), trace | 0 | 0 | 2 | 1
  Occult Blood, 24 hours post-dose (Day 1), 1+ | 1 | 0 | 0 | 0
  Occult Blood, 24 hours post-dose (Day 1), 2+ | 1 | 0 | 0 | 0
  Occult Blood, 24 hours post-dose (Day 1), 3+ | 0 | 0 | 0 | 0
  Glucose, 24 hours post-dose (Day 1), negative | 4 | 5 | 5 | 8
  Glucose, 24 hours post-dose (Day 1), trace | 0 | 0 | 0 | 0
  Glucose, 24 hours post-dose (Day 1), 1+ | 0 | 0 | 0 | 0
  Glucose, 24 hours post-dose (Day 1), 2+ | 0 | 0 | 0 | 0
  Glucose, 24 hours post-dose (Day 1), 3+ | 0 | 0 | 1 | 0
  Ketones, 24 hours post-dose (Day 1), negative | 4 | 4 | 3 | 8
  Ketones, 24 hours post-dose (Day 1), trace | 0 | 1 | 3 | 0
  Ketones, 24 hours post-dose (Day 1), 1+ | 0 | 0 | 0 | 0
  Ketones, 24 hours post-dose (Day 1), 2+ | 0 | 0 | 0 | 0
  Ketones, 24 hours post-dose (Day 1), 3+ | 0 | 0 | 0 | 0
  Protein, 24 hours post-dose (Day 1), negative | 4 | 4 | 6 | 8
  Protein, 24 hours post-dose (Day 1), trace | 0 | 1 | 0 | 0
  Protein, 24 hours post-dose (Day 1), 1+ | 0 | 0 | 0 | 0
  Protein, 24 hours post-dose (Day 1), 2+ | 0 | 0 | 0 | 0
  Protein, 24 hours post-dose (Day 1), 3+ | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in supine position after at least a 5-minute rest. Change from Baseline in pulse rate was evaluated. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose); 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours post-dose (Day 1); and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Beats per minute
  0.5 hour post-dose (Day 1), n=4,5,6,8 | -1.3 (5.85) | -0.8 (3.42) | 3.5 (8.64) | 3.6 (6.00)
  1 hour post-dose (Day 1), n=4,5,6,8 | -3.0 (6.98) | 0.8 (6.69) | -0.7 (3.67) | -1.0 (3.93)
  2 hours post-dose (Day 1), n=4,5,6,8 | -5.0 (7.62) | -0.4 (1.95) | -1.8 (6.65) | 1.0 (5.93)
  4 hours post-dose (Day 1), n=4,5,6,8 | -1.8 (6.80) | 11.6 (13.67) | -1.2 (6.40) | -0.8 (7.42)
  8 hours post-dose (Day 1), n=4,4,6,8: number analyzed (Participants) | 4 | 4 | 6 | 8
  8 hours post-dose (Day 1), n=4,4,6,8 | 2.8 (6.90) | 1.8 (5.19) | 5.7 (5.85) | 8.6 (9.83)
  24 hours post-dose (Day 1), n=4,5,6,8 | 4.3 (11.27) | 3.6 (6.50) | 7.5 (7.12) | 13.0 (9.20)
  Day 7 to Day 14, n=4,5,6,8 | 10.0 (14.31) | 4.4 (5.86) | 5.3 (6.25) | 9.8 (8.36)

19. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in supine position after at least a 5-minute rest. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose); 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours and 24 hours post-dose (Day 1); and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Breaths per minute
  0.5 hour post-dose (Day 1), n=4,5,6,8 | -2.5 (3.11) | -3.4 (4.39) | -2.2 (4.92) | 0.1 (1.13)
  1 hour post-dose (Day 1), n=4,5,6,8 | -2.8 (1.71) | -3.2 (5.67) | 1.8 (9.22) | 0.0 (0.76)
  2 hours post-dose (Day 1), n=4,5,6,8 | -2.0 (2.16) | -2.6 (2.97) | -3.0 (4.52) | -1.0 (4.50)
  4 hours post-dose (Day 1), n=4,5,6,8 | -2.5 (2.08) | -2.2 (5.63) | -2.2 (3.54) | 0.1 (0.64)
  8 hours post-dose (Day 1), n=4,4,6,8: number analyzed (Participants) | 4 | 4 | 6 | 8
  8 hours post-dose (Day 1), n=4,4,6,8 | -2.0 (1.63) | -0.3 (3.50) | 0.2 (2.56) | 1.1 (2.59)
  24 hours post-dose (Day 1), n=4,5,6,8 | -1.8 (0.96) | 0.8 (2.28) | 0.3 (2.58) | -0.1 (1.81)
  Day 7 to Day 14, n=4,5,6,8 | -0.5 (1.73) | -0.4 (3.58) | 2.0 (2.28) | 0.3 (1.16)

20. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in supine position after at least a 5-minute rest. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Millimeters of mercury
  DBP, 0.5 hour post-dose (Day 1), n=4,5,6,8 | -3.5 (8.58) | -1.0 (10.42) | -5.0 (14.67) | -3.3 (4.53)
  DBP, 1 hour post-dose (Day 1), n=4,5,6,8 | -2.0 (6.22) | 0.6 (8.56) | -4.3 (9.73) | -2.3 (3.73)
  DBP, 2 hours post-dose (Day 1), n=4,5,6,8 | 0.5 (12.40) | 1.2 (10.55) | -5.8 (8.80) | 3.3 (5.87)
  DBP, 4 hours post-dose (Day 1), n=4,5,6,8 | -1.5 (2.65) | 3.0 (8.37) | -2.7 (13.22) | 1.6 (6.07)
  DBP, 8 hours post-dose (Day 1), n=4,4,6,8: number analyzed (Participants) | 4 | 4 | 6 | 8
  DBP, 8 hours post-dose (Day 1), n=4,4,6,8 | -12.3 (6.65) | -6.3 (8.66) | -10.2 (9.15) | -1.0 (9.32)
  DBP, 24 hours post-dose (Day 1), n=4,5,6,8 | -7.5 (7.94) | -8.6 (9.61) | -2.8 (10.61) | -3.1 (8.46)
  DBP, Day 7 to Day 14, n=4,5,6,8 | -4.5 (7.19) | -2.2 (6.91) | -2.5 (11.78) | 2.8 (12.83)
  SBP, 0.5 hour post-dose (Day 1), n=4,5,6,8 | -2.3 (12.28) | -0.2 (12.60) | -5.2 (6.11) | -0.1 (5.03)
  SBP, 1 hour post-dose (Day 1), n=4,5,6,8 | -1.8 (9.91) | 3.4 (12.68) | -2.7 (9.37) | 3.0 (8.07)
  SBP, 2 hours post-dose (Day 1), n=4,5,6,8 | 1.0 (15.12) | 2.0 (10.20) | -0.7 (18.84) | 2.0 (11.80)
  SBP, 4 hours post-dose (Day 1), n=4,5,6,8 | 5.5 (19.69) | 4.2 (9.34) | 6.3 (13.03) | 6.1 (13.53)
  SBP, 8 hours post-dose (Day 1), n=4,4,6,8: number analyzed (Participants) | 4 | 4 | 6 | 8
  SBP, 8 hours post-dose (Day 1), n=4,4,6,8 | -4.5 (10.38) | 3.0 (16.57) | -5.2 (7.63) | -4.8 (9.65)
  SBP, 24 hours post-dose (Day 1), n=4,5,6,8 | -2.5 (4.51) | -0.2 (14.72) | -4.7 (11.41) | -3.8 (14.85)
  SBP, Day 7 to Day 14, n=4,5,6,8 | 2.0 (21.37) | 6.0 (6.78) | -5.8 (15.07) | -2.1 (9.63)

21. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECGs were obtained at each time point using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and Corrected QT (QTc) intervals. Only those participants who had any abnormal ECG findings are presented. Abnormal ECG findings were categorized as clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: 4 hours and 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Participants
  Abnormal NCS, 4 hours post-dose (Day 1), n=4,5,6,8 | 1 | 3 | 3 | 7
  Abnormal CS, 4 hours post-dose (Day 1), n=4,5,6,8 | 0 | 0 | 0 | 0
  Abnormal NCS, 24 hours post-dose(Day 1), n=3,5,6,8: number analyzed (Participants) | 3 | 5 | 6 | 8
  Abnormal NCS, 24 hours post-dose(Day 1), n=3,5,6,8 | 1 | 3 | 4 | 5
  Abnormal CS, 24 hours post-dose (Day 1), n=3,5,6,8: number analyzed (Participants) | 3 | 5 | 6 | 8
  Abnormal CS, 24 hours post-dose (Day 1), n=3,5,6,8 | 0 | 0 | 0 | 0
  Abnormal NCS, Day 7 to Day 14, n=4,5,6,8 | 1 | 3 | 3 | 3
  Abnormal CS, Day 7 to Day 14, n=4,5,6,8 | 0 | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Pulse Oximetry Parameter: Percent Oxygen in Blood
Description: Percent oxygen in blood was measured using pulse oximetry after the participant had rested for at least 5 minutes. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of oxygen in blood
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Percentage of oxygen in blood
  0.5 hour post-dose (Day 1), n=4,5,6,8 | -1.0 (2.30) | -1.7 (2.77) | 0.8 (2.31) | -0.5 (2.03)
  1 hour post-dose (Day 1), n=4,5,6,8 | -0.7 (2.87) | -2.1 (2.79) | -0.3 (1.03) | -0.9 (2.48)
  2 hours post-dose (Day 1), n=4,5,6,8 | -1.5 (1.91) | -0.7 (1.99) | 0.6 (1.21) | 0.9 (1.37)
  4 hours post-dose (Day 1), n=4,5,6,8 | -0.7 (2.21) | -1.0 (1.87) | -0.3 (1.96) | 0.5 (2.13)
  8 hours post-dose (Day 1), n=4,4,6,8: number analyzed (Participants) | 4 | 4 | 6 | 8
  8 hours post-dose (Day 1), n=4,4,6,8 | -0.7 (2.50) | -0.2 (3.58) | 0.8 (2.31) | 0.4 (2.98)
  24 hours post-dose (Day 1), n=4,5,6,8 | -1.0 (2.00) | -2.3 (3.06) | 2.1 (1.60) | 1.0 (3.28)
  Day 7 to Day 14, n=4,5,6,8 | -0.2 (0.95) | -2.9 (2.37) | 0.5 (3.33) | 0.8 (2.49)

23. Secondary Outcome: Number of Participants With Positive Immunogenicity Results
Description: Immunogenicity samples were collected into a serum-separating tube, mixed by gentle inversion 5 times and left to coagulate at room temperature for a minimum of 30 minutes and a maximum of 60 minutes. All samples were first tested for anti-angiotensin converting enzyme type 2 (ACE2) binding antibodies by screening and confirmation assay steps. If post-dose samples were found to be positive for anti-ACE2 binding antibodies, they would have been further characterized for anti-ACE2 neutralizing antibodies. Number of participants with positive immunogenicity results post-dosing are presented.
Time Frame: Up to Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Participants | 0 | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in Systemic Renin-Angiotensin System (RAS) Peptides: Angiotensin II, Angiotensin (1-5) and Angiotensin (1-7)
Description: Blood samples were collected to evaluate systemic RAS peptides: Angiotensin (Ang) II, Ang (1-7) and Ang (1-5). Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: Baseline (Day 1, Pre-dose); 0.08 hour, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours and 24 hours post-dose (Day 1); and one sample between Day 7 to Day 14 (follow up visit)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  Ang II, 0.08 hour post-dose (Day 1), n=4,5,5,8 | 0.143 [0.028 to 0.723] | 0.185 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75 percentage (%) of the values were below lower limit of quantification. | 1.020 [0.063 to 16.661] | 0.254 [0.078 to 0.831]
  Ang II, 0.5 hour post-dose (Day 1), n=4,5,5,8 | 0.179 [0.040 to 0.792] | 0.210 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.500 [0.065 to 3.825] | 0.211 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang II, 1 hour post-dose (Day 1), n=4,5,5,8 | 0.238 [0.097 to 0.582] | 0.162 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.420 [0.086 to 2.062] | 0.235 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang II, 2 hours post-dose (Day 1), n=4,5,5,8 | 0.230 [0.041 to 1.280] | 0.166 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.393 [0.159 to 0.970] | 0.211 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang II, 4 hours post-dose (Day 1), n=4,5,5,8 | 0.372 [0.159 to 0.872] | 0.187 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.398 [0.161 to 0.980] | 0.387 [0.160 to 0.933]
  Ang II, 8 hours post-dose (Day 1), n=4,5,5,8 | 0.889 [0.148 to 5.327] | 0.669 [0.249 to 1.798] | 0.503 [0.311 to 0.813] | 0.277 [0.080 to 0.963]
  Ang II, 24 hours post-dose (Day 1), n=4,5,5,8 | 2.329 [0.692 to 7.836] | 1.372 [0.462 to 4.070] | 0.763 [0.267 to 2.184] | 0.939 [0.186 to 4.751]
  Ang II, Day 7 to Day 14, n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang II, Day 7 to Day 14, n=4,5,5,7 | 1.625 [0.084 to 31.300] | 2.380 [0.703 to 8.063] | 0.616 [0.115 to 3.307] | 1.826 [0.399 to 8.354]
  Ang (1-5), 0.08 hour post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 0.08 hour post-dose (Day 1), n=4,5,4,6 | 1.884 [0.505 to 7.026] | 4.696 [1.303 to 16.923] | 2.222 [0.774 to 6.373] | 2.982 [1.360 to 6.535]
  Ang (1-5), 0.5 hour post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 0.5 hour post-dose (Day 1), n=4,5,4,6 | 2.342 [0.435 to 12.622] | 5.325 [1.427 to 19.873] | 2.895 [1.206 to 6.950] | 3.187 [1.303 to 7.797]
  Ang (1-5), 1 hour post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 1 hour post-dose (Day 1), n=4,5,4,6 | 2.427 [0.414 to 14.225] | 4.263 [1.463 to 12.418] | 2.572 [0.775 to 8.539] | 3.264 [1.134 to 9.396]
  Ang (1-5), 2 hours post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 2 hours post-dose (Day 1), n=4,5,4,6 | 2.269 [0.344 to 14.945] | 3.499 [1.377 to 8.890] | 3.423 [0.698 to 16.789] | 2.463 [0.982 to 6.174]
  Ang (1-5), 4 hours post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 4 hours post-dose (Day 1), n=4,5,4,6 | 2.442 [0.344 to 17.340] | 2.740 [1.245 to 6.033] | 3.513 [0.750 to 16.459] | 2.717 [1.033 to 7.146]
  Ang (1-5), 8 hours post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 8 hours post-dose (Day 1), n=4,5,4,6 | 4.365 [1.094 to 17.420] | 4.125 [0.716 to 23.775] | 6.691 [0.812 to 55.117] | 4.882 [1.581 to 15.072]
  Ang (1-5), 24 hours post-dose (Day 1), n=4,5,4,6: number analyzed (Participants) | 4 | 5 | 4 | 6
  Ang (1-5), 24 hours post-dose (Day 1), n=4,5,4,6 | 2.397 [0.879 to 6.536] | 3.701 [1.413 to 9.690] | 2.573 [0.403 to 16.426] | 5.117 [1.910 to 13.712]
  Ang (1-5), Day 7 to Day 14, n=4,5,3,6: number analyzed (Participants) | 4 | 5 | 3 | 6
  Ang (1-5), Day 7 to Day 14, n=4,5,3,6 | 1.469 [0.714 to 3.020] | 2.110 [0.775 to 5.744] | 0.548 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.642 [0.781 to 3.450]
  Ang (1-7), 0.08 hour post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 0.08 hour post-dose (Day 1), n=4,5,5,7 | 2.252 [0.366 to 13.855] | 4.392 [1.405 to 13.732] | 3.465 [1.025 to 11.719] | 1.817 [0.969 to 3.405]
  Ang (1-7), 0.5 hour post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 0.5 hour post-dose (Day 1), n=4,5,5,7 | 2.943 [0.335 to 25.843] | 4.935 [1.383 to 17.617] | 2.242 [0.639 to 7.865] | 2.205 [1.260 to 3.859]
  Ang (1-7), 1 hour post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 1 hour post-dose (Day 1), n=4,5,5,7 | 3.002 [0.318 to 28.319] | 3.494 [1.438 to 8.490] | 2.362 [0.542 to 10.291] | 1.780 [0.783 to 4.047]
  Ang (1-7), 2 hours post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 2 hours post-dose (Day 1), n=4,5,5,7 | 2.311 [0.161 to 33.222] | 4.025 [1.393 to 11.630] | 3.471 [0.651 to 18.500] | 1.949 [1.012 to 3.756]
  Ang (1-7), 4 hours post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 4 hours post-dose (Day 1), n=4,5,5,7 | 3.350 [0.230 to 48.748] | 3.115 [1.349 to 7.190] | 3.623 [0.679 to 19.331] | 1.818 [0.715 to 4.623]
  Ang (1-7), 8 hours post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 8 hours post-dose (Day 1), n=4,5,5,7 | 4.910 [0.654 to 36.845] | 3.517 [0.635 to 19.477] | 6.002 [0.762 to 47.289] | 4.229 [1.433 to 12.477]
  Ang (1-7), 24 hours post-dose (Day 1), n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Ang (1-7), 24 hours post-dose (Day 1), n=4,5,5,7 | 3.423 [0.618 to 18.944] | 4.096 [1.430 to 11.730] | 2.812 [0.503 to 15.732] | 7.095 [2.426 to 20.752]
  Ang (1-7), Day 7 to Day 14, n=4,5,5,6: number analyzed (Participants) | 4 | 5 | 5 | 6
  Ang (1-7), Day 7 to Day 14, n=4,5,5,6 | 1.190 [0.684 to 2.073] | 1.904 [0.596 to 6.089] | 0.925 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.932 [1.111 to 3.362]

25. Secondary Outcome: Change From Baseline in Pulmonary Wedge RAS Peptides: Angiotensin II, Angiotensin (1-5) and Angiotensin (1-7)
Description: Blood samples were collected to evaluate pulmonary wedge RAS peptides: Ang II, Ang (1-5) and Ang (1-7). Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 8
Ratio
  Ang II, 1 hour post-dose (Day 1), n=4,4,4,8 | 0.270 [0.059 to 1.244] | 0.190 [0.025 to 1.475] | 0.394 [0.046 to 3.414] | 0.369 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang II, 2 hours post-dose (Day 1), n=4,4,4,8 | 0.310 [0.068 to 1.419] | 0.193 [0.025 to 1.476] | 0.505 [0.147 to 1.738] | 0.369 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang II, 4 hours post-dose (Day 1), n=4,4,3,8: number analyzed (Participants) | 4 | 4 | 3 | 8
  Ang II, 4 hours post-dose (Day 1), n=4,4,3,8 | 0.332 [0.089 to 1.240] | 0.191 [0.025 to 1.475] | 0.183 [0.038 to 0.879] | 0.420 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  Ang (1-5), 1 hour post-dose (Day 1), n=4,4,4,7: number analyzed (Participants) | 4 | 4 | 4 | 7
  Ang (1-5), 1 hour post-dose (Day 1), n=4,4,4,7 | 2.985 [0.279 to 31.931] | 3.313 [0.892 to 12.310] | 2.709 [0.792 to 9.269] | 1.834 [0.743 to 4.528]
  Ang (1-5), 2 hours post-dose (Day 1), n=4,4,3,7: number analyzed (Participants) | 4 | 4 | 3 | 7
  Ang (1-5), 2 hours post-dose (Day 1), n=4,4,3,7 | 3.443 [0.282 to 42.025] | 4.621 [0.803 to 26.600] | 5.246 [1.386 to 19.859] | 1.562 [0.566 to 4.312]
  Ang (1-5), 4 hours post-dose (Day 1), n=4,4,3,7: number analyzed (Participants) | 4 | 4 | 3 | 7
  Ang (1-5), 4 hours post-dose (Day 1), n=4,4,3,7 | 2.373 [0.401 to 14.050] | 3.213 [0.757 to 13.646] | 5.239 [1.565 to 17.541] | 1.472 [0.575 to 3.768]
  Ang (1-7), 1 hour post-dose (Day 1), n=4,4,4,8 | 2.840 [0.353 to 22.846] | 4.150 [0.912 to 18.880] | 2.993 [0.356 to 25.136] | 1.558 [0.969 to 2.504]
  Ang (1-7), 2 hours post-dose (Day 1), n=4,4,4,8 | 3.376 [0.279 to 40.910] | 3.792 [0.878 to 16.368] | 4.476 [0.612 to 32.754] | 1.589 [0.830 to 3.043]
  Ang (1-7), 4 hours post-dose (Day 1), n=4,4,3,8: number analyzed (Participants) | 4 | 4 | 3 | 8
  Ang (1-7), 4 hours post-dose (Day 1), n=4,4,3,8 | 2.857 [0.362 to 22.550] | 3.151 [0.849 to 11.693] | 8.521 [0.733 to 99.048] | 1.693 [0.818 to 3.504]

26. Secondary Outcome: Systemic RAS Peptide: Angiotensin II/Angiotensin (1-7) Ratio at Indicated Time Points
Description: Blood samples were collected to assess systemic RAS peptides: Angiotensin II and Angiotensin (1-7). Data for angiotensin II/angiotensin (1-7) ratio is presented. Assessment of follow up visit was conducted between any day of Days 7 to 14.
Time Frame: 0.08 hour, 0.5 hour, 1 hour, 2 hours, 4 hours, 8 hours and 24 hours post-dose (Day 1) and one sample between Day 7 to Day 14 (follow up visit)
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  0.08 hour post-dose (Day 1), n=4,5,5,8 | 0.752 [0.175 to 3.239] | 0.463 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.450 [0.313 to 6.711] | 0.843 [0.491 to 1.447]
  0.5 hour post-dose (Day 1), n=4,5,5,8 | 0.718 [0.186 to 2.779] | 0.468 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.097 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.590 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  1 hour post-dose (Day 1), n=4,5,5,8 | 0.937 [0.351 to 2.504] | 0.509 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.875 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.794 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  2 hours post-dose (Day 1), n=4,5,5,8 | 1.174 [0.539 to 2.559] | 0.455 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.558 [0.150 to 2.077] | 0.657 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  4 hours post-dose (Day 1), n=4,5,5,8 | 1.312 [0.571 to 3.011] | 0.659 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 0.540 [0.136 to 2.144] | 1.283 [0.530 to 3.102]
  8 hours post-dose (Day 1), n=4,5,5,8 | 2.139 [0.623 to 7.339] | 2.093 [0.778 to 5.625] | 0.412 [0.083 to 2.055] | 0.439 [0.181 to 1.062]
  24 hours post-dose (Day 1), n=4,5,5,8 | 8.041 [2.416 to 26.757] | 3.682 [1.929 to 7.030] | 1.335 [0.908 to 1.965] | 0.946 [0.435 to 2.054]
  Day 7 to Day 14, n=4,5,5,7: number analyzed (Participants) | 4 | 5 | 5 | 7
  Day 7 to Day 14, n=4,5,5,7 | 16.132 [1.204 to 216.087] | 13.742 [3.829 to 49.326] | 3.278 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 6.156 [2.618 to 14.479]

27. Secondary Outcome: Pulmonary Wedge RAS Peptide: Angiotensin II/Angiotensin (1-7) Ratio at Indicated Time Points
Description: Blood samples were collected to assess pulmonary wedge RAS peptides: Angiotensin II and Angiotensin (1-7). Data for angiotensin II/angiotensin (1-7) ratio is presented.
Time Frame: 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 8
Ratio
  1 hour post-dose (Day 1), n=4,4,4,8 | 0.888 [0.275 to 2.866] | 0.443 [0.108 to 1.821] | 0.620 [0.058 to 6.650] | 0.789 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  2 hours post-dose (Day 1), n=4,4,4,8 | 0.858 [0.253 to 2.908] | 0.493 [0.116 to 2.096] | 0.531 [0.117 to 2.403] | 0.774 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.
  4 hours post-dose (Day 1), n=4,4,3,8: number analyzed (Participants) | 4 | 4 | 3 | 8
  4 hours post-dose (Day 1), n=4,4,3,8 | 1.085 [0.478 to 2.462] | 0.587 [0.172 to 2.003] | 0.148 [0.012 to 1.759] | 0.826 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.

28. Secondary Outcome: Change From Baseline in Disease Biomarkers: N-terminal Pro B-type Natriuretic Peptide (NT Pro-BNP)
Description: Blood samples were collected at specific time points to evaluate NT pro-BNP, a biomarker of disease activity. NT-pro-BNP is a biomarker of cardiac stress or ventricular workload and decreases as a result of reduced force of contraction if pulmonary blood pressure is reduced. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 2 hours, 4 hours and 24 hours post-dose (Day 1)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 4 | 8
Ratio
  2 hours post-dose (Day 1) | 1.034 [0.955 to 1.119] | 1.005 [0.842 to 1.199] | 0.923 [0.795 to 1.071] | 1.015 [0.841 to 1.224]
  4 hours post-dose (Day 1) | 1.025 [0.924 to 1.138] | 1.042 [0.852 to 1.276] | 0.944 [0.795 to 1.120] | 1.074 [0.840 to 1.373]
  24 hours post-dose (Day 1) | 0.606 [0.253 to 1.453] | 0.896 [0.481 to 1.670] | 0.703 [0.430 to 1.151] | 0.810 [0.539 to 1.217]

29. Secondary Outcome: Change From Baseline in Nitrite, Nitrate and Endogenous Nitrite (Biomarkers of Nitric Oxide [NO])
Description: Blood samples were collected at specific time points to evaluate levels of nitrite, nitrate and endogenous nitrite (En. nitrite) (biomarkers of NO). Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 2 hours, 4 hours and 24 hours post-dose (Day 1)
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 8
Ratio
  Nitrite, 2 hours post-dose (Day 1), n=4,4,5,8 | 1.246 [0.440 to 3.533] | 1.029 [0.870 to 1.216] | 0.530 [0.145 to 1.931] | 0.858 [0.797 to 0.923]
  Nitrite, 4 hours post-dose (Day 1), n=4,4,5,8 | 0.760 [0.635 to 0.910] | 0.992 [0.749 to 1.312] | 0.679 [0.420 to 1.096] | 0.770 [0.654 to 0.907]
  Nitrite, 24 hours post-dose (Day 1), n=4,4,4,7: number analyzed (Participants) | 4 | 4 | 4 | 7
  Nitrite, 24 hours post-dose (Day 1), n=4,4,4,7 | 1.038 [0.898 to 1.199] | 1.146 [1.044 to 1.259] | 0.667 [0.245 to 1.814] | 0.914 [0.605 to 1.381]
  Nitrate, 2 hours post-dose (Day 1), n=4,4,5,8 | 1.251 [0.432 to 3.623] | 1.025 [0.862 to 1.218] | 0.485 [0.108 to 2.177] | 0.836 [0.768 to 0.910]
  Nitrate, 4 hours post-dose (Day 1), n=4,4,5,8 | 0.739 [0.595 to 0.917] | 0.977 [0.700 to 1.362] | 0.655 [0.395 to 1.086] | 0.762 [0.649 to 0.895]
  Nitrate, 24 hours post-dose (Day 1), n=4,4,4,7: number analyzed (Participants) | 4 | 4 | 4 | 7
  Nitrate, 24 hours post-dose (Day 1), n=4,4,4,7 | 1.017 [0.853 to 1.212] | 1.149 [1.049 to 1.259] | 0.641 [0.222 to 1.854] | 0.911 [0.597 to 1.390]
  En. nitrite, 2 hours post-dose (Day 1), n=4,4,5,8 | 1.099 [0.798 to 1.512] | 2.036 [0.309 to 13.411] | 1.171 [0.878 to 1.563] | 0.975 [0.647 to 1.469]
  En. nitrite, 4 hours post-dose (Day 1), n=4,4,5,8 | 1.245 [0.665 to 2.330] | 2.819 [0.079 to 100.021] | 1.329 [0.643 to 2.747] | 0.820 [0.466 to 1.443]
  En. nitrite, 24 hours post-dose (Day 1), n=4,4,4,7: number analyzed (Participants) | 4 | 4 | 4 | 7
  En. nitrite, 24 hours post-dose (Day 1), n=4,4,4,7 | 1.290 [0.543 to 3.063] | 1.399 [0.503 to 3.894] | 1.289 [0.501 to 3.316] | 1.271 [0.614 to 2.634]

30. Secondary Outcome: Change From Baseline in Disease Biomarker: Cardiac Troponin-I
Description: Blood samples were collected at specific time points to assess cardiac troponin I. Cardiac troponin I is a biomarker of cardiac stress. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 2 hours, 4 hours and 24 hours post-dose (Day 1)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  2 hours post-dose (Day 1) | 1.565 [0.660 to 3.714] | 1.320 [0.824 to 2.114] | 1.585 [0.657 to 3.822] | 1.414 [0.761 to 2.628]
  4 hours post-dose (Day 1) | 1.968 [0.543 to 7.131] | 1.149 [0.782 to 1.688] | 1.695 [0.592 to 4.856] | 2.030 [1.064 to 3.873]
  24 hours post-dose (Day 1) | 1.316 [0.549 to 3.154] | 1.000 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.000 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification. | 1.000 [NA to NA] — NA indicates confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification.

31. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of Cmax. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic population comprised of participants in the Safety Population for whom a pharmacokinetic sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Micrograms per milliliter | 1.5159 (37.0) | 4.0229 (37.4) | 8.9701 (26.1) | 14.8042 (33.1)

32. Secondary Outcome: Time to Cmax (Tmax) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of tmax. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hours | 0.08333 [0.0833 to 0.1333] | 0.16667 [0.0667 to 0.5000] | 0.10000 [0.0667 to 0.5500] | 0.13333 [0.0833 to 0.6333]

33. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of AUC(0-t). Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hours*micrograms per milliliter | 3.941 (53.6) | 17.874 (30.9) | 46.789 (16.3) | 68.042 (37.0)

34. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of AUC(0-inf). Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 2 | 6 | 7
Hours*micrograms per milliliter | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile for any participants in the 0.1 mg/kg treatment group over the study period; hence, AUC(0-inf) could not be estimated. | 25.26 (7.7) | 52.46 (20.0) | 76.87 (42.1)

35. Secondary Outcome: Last Observed Quantifiable Concentration (Ct) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of Ct. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Micrograms per milliliter | 0.2563 (22.8) | 0.3327 (54.4) | 0.4800 (44.9) | 0.6380 (54.9)

36. Secondary Outcome: Time of the Last Quantifiable Concentration (Tlast) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of tlast. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 6 | 8
Hours | 8.000 [4.20 to 8.47] | 24.000 [8.18 to 24.25] | 24.017 [23.73 to 24.15] | 24.117 [23.97 to 24.28]

37. Secondary Outcome: Plasma Clearance (CL) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of CL. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 2 | 6 | 7
Liters per hour | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile for any participants in the 0.1 mg/kg treatment group over the study period; hence, plasma clearance could not be estimated. | 0.5838 (10.1) | 0.6207 (16.8) | 0.8170 (30.8)

38. Secondary Outcome: Apparent Volume of Distribution of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of apparent volume of distribution. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 2 | 6 | 7
Liters | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile for any participants in the 0.1 mg/kg treatment group over the study period; hence, apparent volume of distribution could not be estimated. | 6.443 (2.4) | 6.593 (20.5) | 8.084 (20.6)

39. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of GSK2586881
Description: Blood samples were collected at indicated time points for evaluation of t1/2. Pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (Day 1) and 0.08, 0.5, 1, 2, 4, 8 and 24 hours post-dose (Day 1)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 2 | 6 | 7
Hours | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile for any participants in the 0.1 mg/kg treatment group over the study period; hence, t1/2 could not be estimated. | 7.651 (7.7) | 7.362 (23.2) | 6.858 (19.6)

40. Other Pre Specified Outcome: Change From Baseline in Cardiac Index (CI)
Description: Cardiac index (CI) was measured using thermodilution. Baseline was defined as the latest pre-dose assessment (Day 1) with a non-missing value, including those from unscheduled visits. Change from Baseline was measured as ratio of post-dose visit value to Baseline value.
Time Frame: Baseline (Day 1, Pre-dose); 1 hour, 2 hours and 4 hours post-dose (Day 1)
Population: Evaluable Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5 | 5 | 8
Ratio
  1 hour post-dose (Day 1) | 1.045 [0.874 to 1.248] | 1.076 [0.947 to 1.223] | 1.084 [0.766 to 1.533] | 0.990 [0.948 to 1.034]
  2 hours post-dose (Day 1) | 1.021 [0.816 to 1.278] | 1.029 [0.951 to 1.113] | 0.926 [0.719 to 1.193] | 1.020 [0.948 to 1.097]
  4 hours post-dose (Day 1) | 1.107 [0.801 to 1.530] | 1.128 [0.941 to 1.352] | 0.889 [0.740 to 1.068] | 1.000 [0.933 to 1.072]

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were reported from start of study treatment and up to Day 28
Description: Non-SAEs and SAEs were reported for Safety Population. Adverse events were presented treatment-wise.
Arm/Group | GSK2586881 0.1 mg/kg | GSK2586881 0.2 mg/kg | GSK2586881 0.4 mg/kg | GSK2586881 0.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/4 | 3/5 | 5/6 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2586881 0.1 mg/kg (N=4) | GSK2586881 0.2 mg/kg (N=5) | GSK2586881 0.4 mg/kg (N=6) | GSK2586881 0.8 mg/kg (N=8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03177603/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03177603/SAP_001.pdf